CLINICAL TRIAL: NCT02083718
Title: G-CSF Mobilized Peripheral Blood Stem Cell Combined With Mesenchymal Stem Cells for Treatment of Poor Graft Function After Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: Peripheral Blood Stem Cell Combined With Mesenchymal Stem Cells for Treatment of Poor Graft Function
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Academy Military Medical Science, China (Industry); Peking University People's Hospital (Other); Sun Yat-sen University (Other); Guangdong Provincial People's Hospital (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFH-PBSC-MSC-2014
Record Dates: First submitted 2014-03-08; First posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Stem Cell Transplantation, Hematopoietic; Poor Graft Function; Hematological Diseases
Keywords: Poor Graft Function; Peripheral Blood Stem Cell; Mesenchymal Stem Cells; Allogeneic hematopoietic stem cell transplantation
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PBSC & MSCs (Experimental): PBSC will be intravenously infused at a dose of 2×10^8/kg. MSCs will be intravenously infused at a dose of 1×10^6 cells/kg once per week. The vital signs of all patients will be closely monitored during and for 24h after administration.If the NEU and PLT levels do not attain the completely response(CR)standards within 28d, a second course of the same treatment will be given.
  Interventions: Biological: PBSC; Biological: MSCs

INTERVENTIONS:
Biological: PBSC
Biological: MSCs

SUMMARY:
The purpose of this study is to evaluate the utility of treating patients experiencing poor graft function after allogeneic hematopoietic stem cell transplantation with Granulocyte Colony-Stimulating Factor (G-CSF) mobilized peripheral stem cell combined (PBSC) with ex-vivo-expanded BM-drived mesenchymal stem cells from third-party donors. Our first objective was to evaluate the effect of such treatment on poor graft function, and second object was to investigate the safety of such treatment.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation(allo-HSCT) is the only cure for many hematologic diseases. However, poor graft function (PGF) is an important complication after allo-HSCT that occurs in 5-27% of patients, and is associated with considerable mortality related to infections or hemorrhagic complications. Treatment of PGF usually involves the prescription of hematopoietic growth factors such as granulocyte colony-stimulating factor (G-CSF), or second transplantation, but these methods are associated with dismal effect or even a significant risk of graft-versus-host disease (GVHD).

Mesenchymal stem cells (MSCs) are a form of multipotent adult stem cells that can be isolated from bone marrow (BM), adipose tissue, and cord blood. Clinical applications of human MSCs include improving hematopoietic engraftment, preventing and treating graft-versus-host disease after allo-HSCT and so on. Some studies have shown that MSCs combined with PBSC or cord blood could be useful to improve engraftment after HSCT. Several reports suggested MSCs might be effective in the treatment of PGF.

However, the efficacy of MSCs as single-drug treatment for PGF is unsatisfactory in our previous study. Therefore, in the present study, G-CSF mobilized PBSC will be used combined with MSCs in the patients with PGF after allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* A patient age of 14-65 years
* Poor graft function developing after allo-HSCT
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Hematopoietic Recovery | 1 year
  Hematopoietic reconstitution post-transplantation is defined as reconstitution of both neutrophil and platelet numbers. Neutrophil reconstitution is defined as occurring on the first 3 consecutive days with an neutrophil(NEU)>0.5×10^9/L, and platelet (PLT) reconstitution is defined as the first >20×10^9/L for 3 consecutive days.

SECONDARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | up to 1 year
  Adverse Events include infections, GVHD, primary underlying disease relapse and any other side effects. Infections will be mainly focused within the first 100 days after treatment. Side effects of treatment includes acute toxicity and late side effects. Acute toxicity principally involves the heart,live and kidney. Late toxic side effects involves principally the development of secondary tumors and relapse of the primary disease.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, MD., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Sanchez-Guijo FM, Lopez-Villar O, Lopez-Anglada L, Villaron EM, Muntion S, Diez-Campelo M, Perez-Simon JA, San Miguel JF, Caballero D, del Canizo MC. Allogeneic mesenchymal stem cell therapy for refractory cytopenias after hematopoietic stem cell transplantation. Transfusion. 2012 May;52(5):1086-91. doi: 10.1111/j.1537-2995.2011.03400.x. Epub 2011 Oct 24. PMID 22023454
- [Background] Meuleman N, Tondreau T, Ahmad I, Kwan J, Crokaert F, Delforge A, Dorval C, Martiat P, Lewalle P, Lagneaux L, Bron D. Infusion of mesenchymal stromal cells can aid hematopoietic recovery following allogeneic hematopoietic stem cell myeloablative transplant: a pilot study. Stem Cells Dev. 2009 Nov;18(9):1247-52. doi: 10.1089/scd.2009.0029. PMID 19309241